CLINICAL TRIAL: NCT04289792
Title: Chemotherapy-based Split Stereotactic Body Radiation Therapy for Borderline Resectable and Locally Advanced Pancreatic Cancer: Study Protocol of a Prospective, Single-arm Phase II Trial
Brief Title: Split-course SBRT for Borderline Resectable and Locally Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Benhua Xu, Director, Fujian Medical University Union Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: splitPC
Record Dates: First submitted 2020-02-20; First posted 2020-02-28 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT with concurrent chemotherapy (Experimental): SBRT with nab-Paclitaxel plus Gemcitabine (nab-P+Gem) chemotherapy
  Interventions: Drug: nab-Paclitaxel+Gemcitabine; Radiation: split-course SBRT

INTERVENTIONS:
Drug: nab-Paclitaxel+Gemcitabine — Drug: nab-Paclitaxel 125 mg/m2 IV over approximately 30-45 min on Days 1 and 15, followed by gemcitabine 1000 mg/m2 IV infusion over approximately 30 min on Days 1 and 15 of each 28-day cycle for 6 cycles.
Radiation: split-course SBRT — Radiation: During the first 1 and 2 cycles of chemotherapy, SBRT was given as a single irradiation of 10 Gy ⅹ 4 times (Days 2 and 16 of each 28-day cycle).

SUMMARY:
Exploratory assessment of the efficacy and safety of gemcitabine-albumin-based paclitaxel chemotherapy combined with SBRT in the treatment of newly diagnosed borderline resectable and locally advanced unresectable pancreatic cancer patients with sequential investigator selection (IC).

DETAILED DESCRIPTION:
The question of how to administer adequate chemotherapy to synchronize SBRT treatment strategy to maximize the benefits of neoadjuvant therapy for improved prognosis of patients with borderline resectable (BRPC) and locally advanced (LAPC) pancreatic cancer is a challenging and debatable issue. No studies have yet evaluated the efficacy of split-course SBRT as the neoadjuvant chemoradiotherapy regimen. The investigators aimed to study whether neoadjuvant chemotherapy plus split-course SBRT results in better outcomes in BRPC and LAPC patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old and ≤ 70 years old.
* Histologically or cytologically confirmed adenocarcinoma of the pancreas.
* Borderline resectable or locally advanced pancreatic cancer proven by imaging examinations via multidisciplinary approaches according to NCCN guidelines
* No prior chemotherapy or radiotherapy
* ECOG performance status of 0 or 1.
* Without distant metastasis
* The maximum diameter of the tumor must not exceed 5 cm
* Acceptable hematology parameters: a. Absolute neutrophil count (ANC) ≥1500 cell/mm3 b. Platelet count ≥100,000/mm3 c. Hemoglobin (Hgb)≥9 g/dL
* Acceptable blood chemistry levels: a. AST/SGOT and ALT/SGPT≤2.5× upper limit of normal range (ULN) b. Total bilirubin≤1.5 ULN c. Alkaline phosphatase≤2.5× ULN d. Serum albumin>3 g/dL e. Serum creatinine≤1.5 ULN
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.

Exclusion Criteria:

* Age < 18 years old and > 70 years old. Prior anticancer therapy for pancreatic carcinoma.
* Presence of or history of metastatic pancreatic adenocarcinoma.
* Patients who had surgeries, chemotherapy, or other treatments before inclusion.
* Any other malignancy within 5 years prior to enrollment
* History of allergy or hypersensitivity to nab-paclitaxel or gemcitabine or any of their excipients.
* Peripheral sensory neuropathy Grade > 1
* Serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders.
* Pregnant or breast feeding.
* Patients enrolled in other clinical trials or incompliant with regular follow-up
* Unwillingness or inability to comply with study procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2020-05-09 (Actual); Primary Completion 2024-05-09 (Estimated); Study Completion 2025-05-09 (Estimated)

PRIMARY OUTCOMES:
Kaplan-Meier Estimate of Progression-Free Survival (PFS) | From enrollment to 2 years after the end of treatment
  Progression-free Survival (PFS) was defined as the time from the date of the first dose to the date of disease progression or death (by any cause), whichever is earlier. The analysis day was calculated from enrollment date for one participant who was not treated. Participants who have no disease progression or have not died were censored to last tumor assessment date with progression-free.

SECONDARY OUTCOMES:
Kaplan-Meier Estimates for Time to Treatment Failure (TTF) | From enrollment to 2 years after the end of treatment
  TTF was defined as the time after the first dose of study therapy to discontinuation of study therapy due to disease progression, death by any cause, or the start of a new non-protocol-defined anticancer therapy/surgery.
Disease Control Rate (DCR) | From enrollment to 2 years after the end of treatment
  DCR was defined as the percentage of participants with a CR or PR or SD from of date of first treatment to 16 weeks. Tumor assessments after start of non-protocol-defined anticancer therapy were excluded.
Overall Response Rate (ORR) | From enrollment to 2 years after the end of treatment
  ORR was defined as the percentage of participants that achieved a combined incidence of complete (CR) and partial response (PR) using RECIST 1.1 guidelines as assessed by the investigator.
Kaplan-Meier Estimates for Overall Survival (OS) | From enrollment to 2 years after the end of treatment
  Overall survival was defined as the time from the date of first dose of study therapy to the date of death (by any cause).
Participants With Treatment Emergent Adverse Events (TEAEs) | From enrollment to 2 years after the end of treatment
  TEAEs are defined as any adverse event (AE) that begin or worsen on or after the start of study drug or procedure of the study period through the maximum duration of the period plus 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Benhua Xu, PHD, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Saif MW. Pancreatic neoplasm in 2011: an update. JOP. 2011 Jul 8;12(4):316-21. PMID 21737886
- [Background] Oettle H, Neuhaus P, Hochhaus A, Hartmann JT, Gellert K, Ridwelski K, Niedergethmann M, Zulke C, Fahlke J, Arning MB, Sinn M, Hinke A, Riess H. Adjuvant chemotherapy with gemcitabine and long-term outcomes among patients with resected pancreatic cancer: the CONKO-001 randomized trial. JAMA. 2013 Oct 9;310(14):1473-81. doi: 10.1001/jama.2013.279201. PMID 24104372
- [Background] Regine WF, Winter KA, Abrams R, Safran H, Hoffman JP, Konski A, Benson AB, Macdonald JS, Rich TA, Willett CG. Fluorouracil-based chemoradiation with either gemcitabine or fluorouracil chemotherapy after resection of pancreatic adenocarcinoma: 5-year analysis of the U.S. Intergroup/RTOG 9704 phase III trial. Ann Surg Oncol. 2011 May;18(5):1319-26. doi: 10.1245/s10434-011-1630-6. Epub 2011 Mar 10. PMID 21499862
- [Background] Michelakos T, Pergolini I, Castillo CF, Honselmann KC, Cai L, Deshpande V, Wo JY, Ryan DP, Allen JN, Blaszkowsky LS, Clark JW, Murphy JE, Nipp RD, Parikh A, Qadan M, Warshaw AL, Hong TS, Lillemoe KD, Ferrone CR. Predictors of Resectability and Survival in Patients With Borderline and Locally Advanced Pancreatic Cancer who Underwent Neoadjuvant Treatment With FOLFIRINOX. Ann Surg. 2019 Apr;269(4):733-740. doi: 10.1097/SLA.0000000000002600. PMID 29227344
- [Background] Gao S, Zhu X, Shi X, Cao K, Bian Y, Jiang H, Wang K, Guo S, Zhang H, Jin G. Comparisons of different neoadjuvant chemotherapy regimens with or without stereotactic body radiation therapy for borderline resectable pancreatic cancer: study protocol of a prospective, randomized phase II trial (BRPCNCC-1). Radiat Oncol. 2019 Mar 27;14(1):52. doi: 10.1186/s13014-019-1254-8. PMID 30917842
- [Background] Zhong J, Patel K, Switchenko J, Cassidy RJ, Hall WA, Gillespie T, Patel PR, Kooby D, Landry J. Outcomes for patients with locally advanced pancreatic adenocarcinoma treated with stereotactic body radiation therapy versus conventionally fractionated radiation. Cancer. 2017 Sep 15;123(18):3486-3493. doi: 10.1002/cncr.30706. Epub 2017 May 10. PMID 28493288
- [Background] Mellon EA, Hoffe SE, Springett GM, Frakes JM, Strom TJ, Hodul PJ, Malafa MP, Chuong MD, Shridhar R. Long-term outcomes of induction chemotherapy and neoadjuvant stereotactic body radiotherapy for borderline resectable and locally advanced pancreatic adenocarcinoma. Acta Oncol. 2015 Jul;54(7):979-85. doi: 10.3109/0284186X.2015.1004367. Epub 2015 Mar 3. PMID 25734581
- [Background] Chuong MD, Springett GM, Weber J, Klapman J, et al. Induction gemcitabine-based chemotherapy and neoadjuvant stereotactic body radiation therapy achieve high margin-negative resection rates for borderline resectable pancreatic cancer. Journal of Radiation Oncology. 2012;1:273-281
- [Background] Polistina F, Costantin G, Casamassima F, Francescon P, Guglielmi R, Panizzoni G, Febbraro A, Ambrosino G. Unresectable locally advanced pancreatic cancer: a multimodal treatment using neoadjuvant chemoradiotherapy (gemcitabine plus stereotactic radiosurgery) and subsequent surgical exploration. Ann Surg Oncol. 2010 Aug;17(8):2092-101. doi: 10.1245/s10434-010-1019-y. Epub 2010 Mar 12. PMID 20224860
- [Background] Rombouts SJ, Walma MS, Vogel JA, van Rijssen LB, Wilmink JW, Mohammad NH, van Santvoort HC, Molenaar IQ, Besselink MG. Systematic Review of Resection Rates and Clinical Outcomes After FOLFIRINOX-Based Treatment in Patients with Locally Advanced Pancreatic Cancer. Ann Surg Oncol. 2016 Dec;23(13):4352-4360. doi: 10.1245/s10434-016-5373-2. Epub 2016 Jul 1. PMID 27370653
- [Background] Moningi S, Dholakia AS, Raman SP, Blackford A, Cameron JL, Le DT, De Jesus-Acosta AM, Hacker-Prietz A, Rosati LM, Assadi RK, Dipasquale S, Pawlik TM, Zheng L, Weiss MJ, Laheru DA, Wolfgang CL, Herman JM. The Role of Stereotactic Body Radiation Therapy for Pancreatic Cancer: A Single-Institution Experience. Ann Surg Oncol. 2015 Jul;22(7):2352-8. doi: 10.1245/s10434-014-4274-5. Epub 2015 Jan 7. PMID 25564157
- [Background] Herman JM, Chang DT, Goodman KA, Dholakia AS, Raman SP, Hacker-Prietz A, Iacobuzio-Donahue CA, Griffith ME, Pawlik TM, Pai JS, O'Reilly E, Fisher GA, Wild AT, Rosati LM, Zheng L, Wolfgang CL, Laheru DA, Columbo LA, Sugar EA, Koong AC. Phase 2 multi-institutional trial evaluating gemcitabine and stereotactic body radiotherapy for patients with locally advanced unresectable pancreatic adenocarcinoma. Cancer. 2015 Apr 1;121(7):1128-37. doi: 10.1002/cncr.29161. Epub 2014 Dec 23. PMID 25538019
- [Background] Kharofa J, Mierzwa M, Olowokure O, Sussman J, Latif T, Gupta A, Xie C, Patel S, Esslinger H, Mcgill B, Wolf E, Ahmad SA. Pattern of Marginal Local Failure in a Phase II Trial of Neoadjuvant Chemotherapy and Stereotactic Body Radiation Therapy for Resectable and Borderline Resectable Pancreas Cancer. Am J Clin Oncol. 2019 Mar;42(3):247-252. doi: 10.1097/COC.0000000000000518. PMID 30724781
- [Background] Shaib WL, Hawk N, Cassidy RJ, Chen Z, Zhang C, Brutcher E, Kooby D, Maithel SK, Sarmiento JM, Landry J, El-Rayes BF. A Phase 1 Study of Stereotactic Body Radiation Therapy Dose Escalation for Borderline Resectable Pancreatic Cancer After Modified FOLFIRINOX (NCT01446458). Int J Radiat Oncol Biol Phys. 2016 Oct 1;96(2):296-303. doi: 10.1016/j.ijrobp.2016.05.010. Epub 2016 May 24. PMID 27475674
- [Background] Bae SH, Kim MS, Kim SY, Jang WI, Cho CK, Yoo HJ, Kim KB, Lee DH, Han CJ, Yang KY, Kim SB. Severe intestinal toxicity after stereotactic ablative radiotherapy for abdominopelvic malignancies. Int J Colorectal Dis. 2013 Dec;28(12):1707-13. doi: 10.1007/s00384-013-1717-6. Epub 2013 Jun 18. PMID 23775098
- [Background] Rostom AY, Tahir S, Gershuny AR, Kandil A, Folkes A, White WF. Once weekly irradiation for carcinoma of the bladder. Int J Radiat Oncol Biol Phys. 1996 May 1;35(2):289-92. doi: 10.1016/0360-3016(96)00063-6. PMID 8635935
- [Background] McLaren DB, Morrey D, Mason MD. Hypofractionated radiotherapy for muscle invasive bladder cancer in the elderly. Radiother Oncol. 1997 May;43(2):171-4. doi: 10.1016/s0167-8140(97)01943-9. PMID 9192963
- [Background] Scholten AN, Leer JW, Collins CD, Wondergem J, Hermans J, Timothy A. Hypofractionated radiotherapy for invasive bladder cancer. Radiother Oncol. 1997 May;43(2):163-9. doi: 10.1016/s0167-8140(96)01893-2. PMID 9192962
- [Background] Jose CC, Price A, Norman A, Jay G, Huddart R, Dearnaley DP, Horwich A. Hypofractionated radiotherapy for patients with carcinoma of the bladder. Clin Oncol (R Coll Radiol). 1999;11(5):330-3. doi: 10.1053/clon.1999.9075. PMID 10591821
- [Background] Hafeez S, McDonald F, Lalondrelle S, McNair H, Warren-Oseni K, Jones K, Harris V, Taylor H, Khoo V, Thomas K, Hansen V, Dearnaley D, Horwich A, Huddart R. Clinical Outcomes of Image Guided Adaptive Hypofractionated Weekly Radiation Therapy for Bladder Cancer in Patients Unsuitable for Radical Treatment. Int J Radiat Oncol Biol Phys. 2017 May 1;98(1):115-122. doi: 10.1016/j.ijrobp.2017.01.239. Epub 2017 Feb 9. PMID 28586948
- [Background] Bledsoe TJ, Noble AR, Reddy CA, Burkey BB, Greskovich JF, Nwizu T, Adelstein DJ, Saxton JP, Koyfman SA. Split-Course Accelerated Hypofractionated Radiotherapy (SCAHRT): A Safe and Effective Option for Head and Neck Cancer in the Elderly or Infirm. Anticancer Res. 2016 Mar;36(3):933-9. PMID 26976981
- [Background] Suker M, Beumer BR, Sadot E, Marthey L, Faris JE, Mellon EA, El-Rayes BF, Wang-Gillam A, Lacy J, Hosein PJ, Moorcraft SY, Conroy T, Hohla F, Allen P, Taieb J, Hong TS, Shridhar R, Chau I, van Eijck CH, Koerkamp BG. FOLFIRINOX for locally advanced pancreatic cancer: a systematic review and patient-level meta-analysis. Lancet Oncol. 2016 Jun;17(6):801-810. doi: 10.1016/S1470-2045(16)00172-8. Epub 2016 May 6. PMID 27160474
- [Background] Muranaka T, Kuwatani M, Komatsu Y, Sawada K, Nakatsumi H, Kawamoto Y, Yuki S, Kubota Y, Kubo K, Kawahata S, Kawakubo K, Kawakami H, Sakamoto N. Comparison of efficacy and toxicity of FOLFIRINOX and gemcitabine with nab-paclitaxel in unresectable pancreatic cancer. J Gastrointest Oncol. 2017 Jun;8(3):566-571. doi: 10.21037/jgo.2017.02.02. PMID 28736643
- [Background] Verma V, Lazenby AJ, Zheng D, Bhirud AR, Ly QP, Are C, Sasson AR, Lin C. Dosimetric parameters correlate with duodenal histopathologic damage after stereotactic body radiotherapy for pancreatic cancer: Secondary analysis of a prospective clinical trial. Radiother Oncol. 2017 Mar;122(3):464-469. doi: 10.1016/j.radonc.2016.12.030. Epub 2017 Jan 12. PMID 28089484
- [Background] Benedict SH, Yenice KM, Followill D, Galvin JM, Hinson W, Kavanagh B, Keall P, Lovelock M, Meeks S, Papiez L, Purdie T, Sadagopan R, Schell MC, Salter B, Schlesinger DJ, Shiu AS, Solberg T, Song DY, Stieber V, Timmerman R, Tome WA, Verellen D, Wang L, Yin FF. Stereotactic body radiation therapy: the report of AAPM Task Group 101. Med Phys. 2010 Aug;37(8):4078-101. doi: 10.1118/1.3438081. PMID 20879569
- [Background] Blomstrand H, Scheibling U, Bratthall C, Green H, Elander NO. Real world evidence on gemcitabine and nab-paclitaxel combination chemotherapy in advanced pancreatic cancer. BMC Cancer. 2019 Jan 8;19(1):40. doi: 10.1186/s12885-018-5244-2. PMID 30621618
- [Background] Gemenetzis G, Groot VP, Blair AB, Laheru DA, Zheng L, Narang AK, Fishman EK, Hruban RH, Yu J, Burkhart RA, Cameron JL, Weiss MJ, Wolfgang CL, He J. Survival in Locally Advanced Pancreatic Cancer After Neoadjuvant Therapy and Surgical Resection. Ann Surg. 2019 Aug;270(2):340-347. doi: 10.1097/SLA.0000000000002753. PMID 29596120
- [Background] Jang JY, Han Y, Lee H, Kim SW, Kwon W, Lee KH, Oh DY, Chie EK, Lee JM, Heo JS, Park JO, Lim DH, Kim SH, Park SJ, Lee WJ, Koh YH, Park JS, Yoon DS, Lee IJ, Choi SH. Oncological Benefits of Neoadjuvant Chemoradiation With Gemcitabine Versus Upfront Surgery in Patients With Borderline Resectable Pancreatic Cancer: A Prospective, Randomized, Open-label, Multicenter Phase 2/3 Trial. Ann Surg. 2018 Aug;268(2):215-222. doi: 10.1097/SLA.0000000000002705. PMID 29462005
- [Background] Bednar F, Zenati MS, Steve J, Winters S, Ocuin LM, Bahary N, Hogg ME, Zeh HJ 3rd, Zureikat AH. Analysis of Predictors of Resection and Survival in Locally Advanced Stage III Pancreatic Cancer: Does the Nature of Chemotherapy Regimen Influence Outcomes? Ann Surg Oncol. 2017 May;24(5):1406-1413. doi: 10.1245/s10434-016-5707-0. Epub 2016 Nov 28. PMID 27896518
- [Background] Conroy T, Bachet JB, Ayav A, Huguet F, Lambert A, Caramella C, Marechal R, Van Laethem JL, Ducreux M. Current standards and new innovative approaches for treatment of pancreatic cancer. Eur J Cancer. 2016 Apr;57:10-22. doi: 10.1016/j.ejca.2015.12.026. Epub 2016 Feb 4. PMID 26851397
- [Background] Murphy JD, Christman-Skieller C, Kim J, Dieterich S, Chang DT, Koong AC. A dosimetric model of duodenal toxicity after stereotactic body radiotherapy for pancreatic cancer. Int J Radiat Oncol Biol Phys. 2010 Dec 1;78(5):1420-6. doi: 10.1016/j.ijrobp.2009.09.075. Epub 2010 Apr 14. PMID 20399033
- [Background] Paik EK, Kim MS, Seo YS, Jang WI, Kang JK, Cho CK, Yoo HJ. Feasibility of split-course stereotactic ablative radiotherapy for oligometastases. Jpn J Clin Oncol. 2018 Jun 1;48(6):548-554. doi: 10.1093/jjco/hyy062. PMID 29722825
- [Background] Gielda BT, Marsh JC, Zusag TW, Faber LP, Liptay M, Basu S, Warren WH, Fidler MJ, Batus M, Abrams RA, Bonomi P. Split-course chemoradiotherapy for locally advanced non-small cell lung cancer: a single-institution experience of 144 patients. J Thorac Oncol. 2011 Jun;6(6):1079-86. doi: 10.1097/JTO.0b013e3182199a7c. PMID 21532501
- [Background] Milas L, Milas MM, Mason KA. Combination of taxanes with radiation: preclinical studies. Semin Radiat Oncol. 1999 Apr;9(2 Suppl 1):12-26. PMID 10210536
- [Background] Milas L, Fujii T, Hunter N, Elshaikh M, Mason K, Plunkett W, Ang KK, Hittelman W. Enhancement of tumor radioresponse in vivo by gemcitabine. Cancer Res. 1999 Jan 1;59(1):107-14. PMID 9892194
- [Background] Higuchi Y, Serizawa T, Nagano O, Matsuda S, Ono J, Sato M, Iwadate Y, Saeki N. Three-staged stereotactic radiotherapy without whole brain irradiation for large metastatic brain tumors. Int J Radiat Oncol Biol Phys. 2009 Aug 1;74(5):1543-8. doi: 10.1016/j.ijrobp.2008.10.035. Epub 2009 Jan 8. PMID 19135317
- [Background] Hsieh CH, Chang HT, Lin SC, Chen YJ, Wang LY, Hsieh YP, Chen CA, Chong NS, Lin SL, Chen CY, Shueng PW. Toxic risk of stereotactic body radiotherapy and concurrent helical tomotherapy followed by erlotinib for non-small-cell lung cancer treatment--case report. BMC Cancer. 2010 Dec 31;10:696. doi: 10.1186/1471-2407-10-696. PMID 21194444
- [Background] Angelov L, Mohammadi AM, Bennett EE, Abbassy M, Elson P, Chao ST, Montgomery JS, Habboub G, Vogelbaum MA, Suh JH, Murphy ES, Ahluwalia MS, Nagel SJ, Barnett GH. Impact of 2-staged stereotactic radiosurgery for treatment of brain metastases >/= 2 cm. J Neurosurg. 2018 Aug;129(2):366-382. doi: 10.3171/2017.3.JNS162532. Epub 2017 Sep 22. PMID 28937324
- [Background] Carlson DJ, Keall PJ, Loo BW Jr, Chen ZJ, Brown JM. Hypofractionation results in reduced tumor cell kill compared to conventional fractionation for tumors with regions of hypoxia. Int J Radiat Oncol Biol Phys. 2011 Mar 15;79(4):1188-95. doi: 10.1016/j.ijrobp.2010.10.007. Epub 2010 Dec 22. PMID 21183291
- [Background] Brown JM, Carlson DJ, Brenner DJ. The tumor radiobiology of SRS and SBRT: are more than the 5 Rs involved? Int J Radiat Oncol Biol Phys. 2014 Feb 1;88(2):254-62. doi: 10.1016/j.ijrobp.2013.07.022. PMID 24411596
- [Background] Park HJ, Griffin RJ, Hui S, Levitt SH, Song CW. Radiation-induced vascular damage in tumors: implications of vascular damage in ablative hypofractionated radiotherapy (SBRT and SRS). Radiat Res. 2012 Mar;177(3):311-27. doi: 10.1667/rr2773.1. Epub 2012 Jan 9. PMID 22229487
- [Background] Finkelstein SE, Timmerman R, McBride WH, Schaue D, Hoffe SE, Mantz CA, Wilson GD. The confluence of stereotactic ablative radiotherapy and tumor immunology. Clin Dev Immunol. 2011;2011:439752. doi: 10.1155/2011/439752. Epub 2011 Nov 15. PMID 22162711
- [Background] Song CW, Kim MS, Cho LC, Dusenbery K, Sperduto PW. Radiobiological basis of SBRT and SRS. Int J Clin Oncol. 2014 Aug;19(4):570-8. doi: 10.1007/s10147-014-0717-z. Epub 2014 Jul 5. PMID 24993673
- [Background] Filatenkov A, Baker J, Mueller AM, Kenkel J, Ahn GO, Dutt S, Zhang N, Kohrt H, Jensen K, Dejbakhsh-Jones S, Shizuru JA, Negrin RN, Engleman EG, Strober S. Ablative Tumor Radiation Can Change the Tumor Immune Cell Microenvironment to Induce Durable Complete Remissions. Clin Cancer Res. 2015 Aug 15;21(16):3727-39. doi: 10.1158/1078-0432.CCR-14-2824. Epub 2015 Apr 13. PMID 25869387
- [Background] Lee Y, Auh SL, Wang Y, Burnette B, Wang Y, Meng Y, Beckett M, Sharma R, Chin R, Tu T, Weichselbaum RR, Fu YX. Therapeutic effects of ablative radiation on local tumor require CD8+ T cells: changing strategies for cancer treatment. Blood. 2009 Jul 16;114(3):589-95. doi: 10.1182/blood-2009-02-206870. Epub 2009 Apr 6. PMID 19349616
- [Background] Lugade AA, Moran JP, Gerber SA, Rose RC, Frelinger JG, Lord EM. Local radiation therapy of B16 melanoma tumors increases the generation of tumor antigen-specific effector cells that traffic to the tumor. J Immunol. 2005 Jun 15;174(12):7516-23. doi: 10.4049/jimmunol.174.12.7516. PMID 15944250
- [Background] Nishikawa H, Sakaguchi S. Regulatory T cells in tumor immunity. Int J Cancer. 2010 Aug 15;127(4):759-67. doi: 10.1002/ijc.25429. PMID 20518016
- [Background] Aryankalayil MJ, Makinde AY, Gameiro SR, Hodge JW, Rivera-Solis PP, Palayoor ST, Ahmed MM, Coleman CN. Defining molecular signature of pro-immunogenic radiotherapy targets in human prostate cancer cells. Radiat Res. 2014 Aug;182(2):139-48. doi: 10.1667/RR13731.1. Epub 2014 Jul 8. PMID 25003313
- [Derived] Zheng R, Wang C, Huang X, Lin Q, Huang D, Li XB, Huang H, Xu B. Chemotherapy-based split stereotactic body radiation therapy for borderline resectable and locally advanced pancreatic cancer: study protocol of a prospective, single-arm phase II trial. BMJ Open. 2020 Nov 5;10(11):e039900. doi: 10.1136/bmjopen-2020-039900. PMID 33154057